CLINICAL TRIAL: NCT00231335
Title: The Efficacy and Safety of Escitalopram Augmentation of Risperidone and Olanzapine in Treatment Resistant Schizophrenia: a Double Blind Placebo Controlled Pilot Study
Brief Title: Efficacy and Safety Study of Escitalopram Augmentation in Treatment Resistant Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Dragan Bugarski-Kirola, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 408-2005
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2006-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; depression; anxiety; negative symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depression; Anxiety Disorders | interventions — Escitalopram

INTERVENTIONS:
Drug: escitalopram

SUMMARY:
A primary hypothesis to be explored here is that, given its pharmacodynamic profile and hypothesized mechanisms associated with schizophrenia, escitalopram will, in comparison to placebo, be effective when added to risperidone or olanzapine treated group in reducing the severity of resistant symptoms, particularly existing subsyndromal anxiety and depression.

DETAILED DESCRIPTION:
The objective of this trial is to determine the efficacy and safety of augmenting risperidone or olanzapine with escitalopram for treatment of symptoms of schizophrenia in patients with incomplete response to adequate trials of either of the two antipsychotic medications. To our knowledge, this is the first double blind randomized study designed to examine the potential augmentation benefit of escitalopram combined with a commonly used atypical agent in chronic schizophrenic patients with incomplete response to risperidone or olanzapine. The current proposal offers the possibility to test the efficacy of augmentation treatment in a controlled fashion with clinical and biological variables used as indicators of response and tolerability. From a broader perspective, it would test the hypothesis of potential validity of SSRI augmentation strategy in treatment of resistant symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM IV criteria for schizophrenia adn schizoaffective disorder and clinically stable on fixed dose of risperidone or olanzapine for at least 6 weeks.
2. Incomplete response to risperidone or olanzapine for at least 6 weeks per subjective report and minimum score on rating instruments (PANSS total >50 at baseline).
3. Current positive and negative symptoms sufficiently severe to require adjuvant treatment despite good compliance and adequate doses of antipsychotic before trial (risperidone 4 to 6mg/day, olanzapine15 to 20mg/day for 4-6 weeks of treatment).
4. Males and females between 18-55 years of age. No restrictions to recruitment based on race.
5. Able to participate fully in the informed consent process or have legal guardian able to participate in the informed consent process. All prospective research subjects will be screened for decisional capacity using the MacArthur Competence Assessment Tool-Research (MacCAT-CR)
6. Educational level of at least 10th grade.
7. Score on at least on PANSS psychosis items (P1,P2,P3,P5,or P6)>4 adn CGI Severity score >4 at point of maximum severity of illness to date or total PANSS score at baseline assessed as moderate (PANSS total >50).

Exclusion Criteria:

1. Meets full DSM-IV criteria for current Major Depressive Disorder, Bipolar Disorder, Anxiety Disorder or any other active disorder on Axis I. Present but not past history of substance abuse is exclusion criterion.
2. Extrapyramidal symptoms as defined by score of 4 or more on Simpson-Angus rating scale.
3. Non-English speaking.
4. Serious unstable medical illness or any acute medical condition.
5. Known allergy to any study medication.
6. Serious suicidal or homicidal risks.
7. Participation in clinical trial of an investigational drug within 30 days of visit 1.
8. Evidence at screening of any medical conditions including but not limited to: infection, electrolyte abnormality, recent physical trauma, malignancy, autoimmune disorders, endocrine diseases and neurological diseases, history of CNS trauma or active seizure disorder requiring medication and known history of mental retardation.
9. Any other condition, which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with participating in or completing the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Reduction of severity of symptoms defined as decrease of >20% from baseline to final evaluation on the PANSS total score.

SECONDARY OUTCOMES:
Changes on depression/anxiety dimensions of PANSS subscales defined as decrease of >20% from baseline to final evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Bugarski-Kirola, MD, Principal Investigator — Emory University